CLINICAL TRIAL: NCT03236454
Title: Effects and Mechanisms of Cognitive Control Training Combined With Transcranial Direct Current Stimulation (tDCS) in Subjective Cognitive Decline.
Brief Title: tDCS-enhanced Working Memory Training in Subjective Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Apl. Prof., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCDStim-1
Record Dates: First submitted 2017-07-27; First posted 2017-08-02 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Subjective Cognitive Decline
Keywords: brain stimulation; cognitive training; cognition; treatment

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sham Stimulation: Ramping up over 50 seconds at the beginning and an equal amount of time for tapering off at the end
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal tDCS (Active Comparator): DC-Stimulator MC, NeuroConn: 20 minutes of 2 mA anodal stimulation
  Interventions: Device: DC-Stimulator MC, NeuroConn
- sham tDCS (Sham Comparator): DC-Stimulator MC, NeuroConn: 20 minutes of sham stimulation; Ramping up over 50 seconds at the beginning and an equal amount of time for tapering off at the end;
  Interventions: Device: DC-Stimulator MC, NeuroConn

INTERVENTIONS:
Device: DC-Stimulator MC, NeuroConn — 20 minutes of 2 mA anodal stimulation; Electrode placement: left dorsolateral prefrontal cortex (F3, EEG 10/20 system), return electrode at the right upper arm.

SUMMARY:
This 2-armed randomized, sham-controlled, single-blind study aims at providing evidence for the efficacy of a transcranial direct current stimulation (tDCS)-enhanced cognitive control training (PASAT) in participants with subjective cognitive decline (SCD). Overall, the study will include 30 participants. Each participant will take part in a four weeks training (12 sessions); 50% of the participants will receive 2mA anodal tDCS for 20 minutes applied to the left dorsolateral prefrontal cortex (dlPFC), the other half will receive sham stimulation. Event-related potentials (ERPs) evoked by the feedback on the correctness of the response at baseline and after training will be measured with EEG as neurophysiological signatures of cognitive control. Near and far transfer will be assessed by a verbal 2-back task and the Trail Making Test A and B. The amount of worrying regarding the memory impairment will be quantified by means of a 10 point Likert-Scale. Together with changes of PASAT performance these measures will be obtained before and after the tDCS-enhanced training. Follow-up assessments 3, 12 and 24 months after training will investigate the stability of training effects.

ELIGIBILITY:
Inclusion Criteria:

Men and women, aged 60 years and above Native German speaker Subjective feeling of worsening cognitive abilities, including memory Present concerns regarding the subjective memory decline Right handedness

Exclusion Criteria:

* Present objective cognitive impairment (Mini-Mental State Examination < 24)
* Current depression or depressive episode (Geriatric Depression Scale > 5)
* Current substance abuse
* Presence of other psychiatric disorders (MINI International Neuropsychiatric Interview)
* History of epilepsy
* Presence of other neurological disorders
* Absence of independent living skills (Instrumental Activities Of Daily Living, IADL) Scale)
* Metallic implants near the electrodes (i.e. pacemakers)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in amount of worrying regarding the memory impairment | 4 weeks
  The amount of worrying regarding the memory impairment will be quantified by means of a 10-point Likert-Scale

SECONDARY OUTCOMES:
Group comparison (active vs. sham tDCS) regarding the change in amount of correct answers in the PASAT task from baseline to end of training period. | 4 weeks
Group comparison (active vs. sham tDCS) regarding the change in amount of correct answers in the verbal 2-back task (pre-session outcomes compared with post-session and follow-up outcomes). | 2 years
Group comparison (active vs. sham tDCS) regarding changes in Trail Making Task A and B outcomes (pre-session outcomes compared with post-session and follow-up outcomes). | 2 years
Group comparison (active vs. sham tDCS) regarding changes in Satisfaction With Life Scale outcomes (pre-session outcomes compared with post-session and follow-up outcomes). | 2 years
Group comparison (active vs. sham tDCS) regarding changes in the Neuropsychological Test Battery CERAD-Plus (pre-session outcomes compared with follow-up outcomes). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, MD, Principal Investigator — University of Tübingen, Department of Psychiatry and Psychotherapy
Locations (1):
- University of Tübingen, Department of Psychiatry and Psychotherapy, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided